CLINICAL TRIAL: NCT00006106
Title: Phase I Study of Intraarterial ONYX-015 in Combination With Intravenous Cisplatin and Fluorouracil in Patients With Advanced Squamous Cell Cancer of the Head and Neck
Brief Title: ONYX-015 With Cisplatin and Fluorouracil in Treating Patients With Advanced Head and Neck Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: Dana-Farber Cancer Institute (Other)
Purpose: Treatment
Other Study IDs: DFCI-98320; CDR0000068117 (Registry Identifier: PDQ (Physician Data Query)); NCI-G00-1832
Record Dates: First submitted 2000-08-03; First posted 2004-04-29 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2006-12

CONDITIONS: Lip and Oral Cavity Cancer; Head and Neck Cancer; Oropharyngeal Cancer
Keywords: adult solid tumor; body system/site cancer; cancer; cellular diagnosis, hypopharyngeal cancer; cellular diagnosis, laryngeal cancer; cellular diagnosis, lip and oral cavity cancer; cellular diagnosis, nasopharyngeal cancer; cellular diagnosis, oropharyngeal cancer; cellular diagnosis, paranasal sinus and nasal cavity cancer; head and neck cancer; hypopharyngeal cancer; hypopharyngeal squamous cell carcinoma; laryngeal cancer; laryngeal squamous cell carcinoma; lip and oral cavity cancer; lip and oral cavity squamous cell carcinoma; metastatic squamous neck cancer with occult primary; nasopharyngeal cancer; nasopharyngeal squamous cell carcinoma; oropharyngeal cancer; oropharyngeal squamous cell carcinoma; paranasal sinus and nasal cavity cancer; paranasal sinus and nasal cavity squamous cell carcinoma; recurrent hypopharyngeal cancer; recurrent laryngeal cancer; recurrent lip and oral cavity cancer; recurrent metastatic squamous neck cancer with occult primary; recurrent nasopharyngeal cancer; recurrent oropharyngeal cancer; recurrent paranasal sinus and nasal cavity cancer; recurrent squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; solid tumor; stage III hypopharyngeal cancer; stage III laryngeal cancer; stage III lip and oral cavity cancer; stage III nasopharyngeal cancer; stage III oropharyngeal cancer; stage III paranasal sinus and nasal cavity cancer; stage III squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV hypopharyngeal cancer; stage IV laryngeal cancer; stage IV lip and oral cavity cancer; stage IV nasopharyngeal cancer; stage IV oropharyngeal cancer; stage IV paranasal sinus and nasal cavity cancer; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; stage, hypopharyngeal cancer; stage, laryngeal cancer; stage, lip and oral cavity cancer; stage, metastatic squamous neck cancer with occult primary; stage, nasopharyngeal cancer; stage, oropharyngeal cancer; stage, paranasal sinus and nasal cavity cancer
MeSH Terms: conditions — Mouth Neoplasms; Head and Neck Neoplasms; Oropharyngeal Neoplasms; Neoplasms; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Lymphoid Interstitial Pneumonia; Nasopharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Fluorouracil; dl1520

INTERVENTIONS:
Drug: cisplatin
Drug: fluorouracil
Drug: ONYX-015

SUMMARY:
RATIONALE: A specially modified virus called ONYX-015 may be able to kill tumor cells while leaving normal cells undamaged. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining ONYX-015 with chemotherapy may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of ONYX-015 combined with cisplatin and fluorouracil in treating patients who have advanced head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the feasibility and maximum tolerated dose (MTD) of intraarterial ONYX-015 in patients with advanced squamous cell cancer of the head and neck.

II. Determine the feasibility and tolerability of intraarterial ONYX-015 at the MTD OR maximum theraputic dose, whichever is lower, in combination with intravenous cisplatin and fluorouracil in these patients.

III. Determine the qualitative distribution of ONYX-015 within a limited tumor biopsy and a normal mucosal biopsy at different dose levels.

IV. Determine the response of these patients to intraarterial ONYX-015. V. Determine the response of these patients to cisplatin and fluorouracil following intraarterial ONYX-015.

PROTOCOL OUTLINE: This is a dose escalation study. Patients receive intraarterial infusions of ONYX-015. Treatment repeats once in 3-4 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-8 patients receive escalating doses of ONYX-015 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 5 patients experience dose limiting toxicity.

Patients in cohorts 1-4 are followed for 5 days after infusion, weekly for 3 weeks, at week 6, and monthly thereafter for 4 months.

A fifth or final cohort of 10 patients will receive ONYX-015 at the MTD. If the MTD was not determined in cohorts 1-4, patients receive the highest dose administered to cohort 4. Beginning 1-2 days after ONYX-015 infusion, patients receive cisplatin IV over 30-60 minutes once and fluorouracil IV continuously over 4 days. Treatment repeats in 4 weeks in the absence of disease progression or unacceptable toxicity. Cisplatin and fluorouracil IV treatment continues every 3-4 weeks at the discretion of the treating oncologist.

Patients in cohort 5 are followed for 5 days after initial infusion, weekly for 4 weeks, at week 8, and monthly thereafter for 4 months.

PROJECTED ACCRUAL:

A total of 23-28 patients will be accrued for this study.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Histologically confirmed squamous cell carcinoma of the head and neck (SCCHN) that is incurable by standard therapy
* Measurable or evaluable disease
* Multiple SCCHN primaries allowed
* Metastases allowed if tumor to be treated is confined to head and neck region

--Prior/Concurrent Therapy--

* Biologic therapy: Recovered from prior biologic therapy
* Chemotherapy: At least 3 weeks since prior chemotherapy and recovered
* Endocrine therapy: Recovered from prior endocrine therapy
* Radiotherapy: At least 12 weeks since prior radiotherapy and recovered
* Surgery: Recovered from prior surgery
* Other: Recovered from any prior diagnostic or theraputic procedures

--Patient Characteristics--

* Age: 18 to physiologic 79
* Performance status: ECOG 0-2
* Life expectancy: Over 3 months
* Hematopoietic: WBC greater than 3,000/mm3 OR Absolute neutrophil count greater than 2,000/mm3; Platelet count greater than 100,000/mm3; Hemoglobin greater than 10 g/dL (transfusions allowed if not used solely to meet eligibility criteria)
* Hepatic: SGOT less than 2.5 times upper limit of normal (ULN); Alkaline phosphatase less than 3 times ULN; Bilirubin no greater than 1.5 times ULN
* Renal: Creatinine less than 1.6 mg/dL OR Creatinine clearance greater than 50 mL/min
* Cardiovascular: No active cardiovascular disease that would limit physical activity (i.e., ability to walk 50 feet without stopping)
* Pulmonary: No active pulmonary disease that would limit physical activity (i.e., ability to walk 50 feet without stopping)
* Other: No other prior or concurrent malignancy within the past 3 years except limited basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix; Adequate and nutritionally balanced enteral intake of at least 1,800 kcal/day (enteral feeding tube dependent allowed); No intravenous alimentation as primary source of calories; No other serious illness or medical condition that would preclude study (i.e., active systemic lupus erythematosus, Crohn's disease or AIDS); No prior immunodeficiency (i.e., HIV infection, organ transplant, or chronic steroid use); Not pregnant or nursing; Negative pregnancy test; Fertile patients must use effective contraception

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 1999-07

CONTACTS AND LOCATIONS:
Overall Officials: Marshall R. Posner, Study Chair — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts